CLINICAL TRIAL: NCT04495608
Title: Multicenter, Double-blind, Placebo-controlled Study to Evaluate the Efficacy and Safety of Fluconazole in Hypercalcicuric Patients With Increased 1.25(OH) 2D Levels
Acronym: FLUCOLITH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 69HCL20_0071; 2020-003011-97 (EudraCT Number)
Record Dates: First submitted 2020-07-23; First posted 2020-08-03 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Nephrolithiasis; Nephrocalcinosis; Hypercalciuria
Keywords: Hypercalciuria; nephrocalcinosis; 1,25-dihydroxyvitamin D; 1-alpha-hydroxylase; fluconazole
MeSH Terms: conditions — Nephrolithiasis; Nephrocalcinosis; Hypercalciuria | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding procedure will be systematic thanks to the indistinguishable nature of the active product and placebo and their packaging.
  Only the biostatistician in charge of the production of the randomization list, the Centre Anti-Poison of Lyon, and the main pharmacy (Pharmacy Department Groupement Hospitalier Centre - Edouard Herriot Hospital - Hospices Civils de Lyon (Lyon, France), responsible for packaging, labeling and dispatching of experimental drugs to the sites, will have access to a decoded list.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fluconazole (Experimental): Fluconazole 50mg capsule (1, 2, 3 or 4 pills to take daily during 18 weeks, corresponding respectively to 50, 100, 150 or 200 mg of fluconazole).
  Interventions: Drug: Fluconazole
- placebo (Placebo Comparator): Placebo (1, 2, 3 or 4 pills to take daily during 18 weeks), same appearance to experimental drug
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fluconazole — Fluconazole 50 mg/capsule or placebo, per os during 18 weeks :
  * From W0 to W2 : 1 caps/ day
  * From W2 to W4 : 1 or 2 caps/day
  * From W4 to W6 : 1, 2 or 3 caps/day
  * From W6 to W18 : 1, 2, 3 or 4 caps/day
  The number of capsules to take will be determined by 24-hours calciuria results performed every 2 weeks during the titration period (W2, W4 and W6).
  During the titration period, if 24-hours calciuria is > 0.1 mmol/kg/day, fluconazole dose will be increased every 2 weeks to 50 mg per intake, with a maximum dose of 200 mg/day. If 24-hour calciuria is ≤ 0.1mmol/kg/day, fluconazole dose will remain stable.
  After W6 and until the end of the study, the treatment dose will remain stable (stable period).
  Arms: fluconazole
Drug: Placebo — Placebo (1, 2, 3 or 4 pills to take daily during 18 weeks), same appearance to experimental drug
  Arms: placebo

SUMMARY:
Hypercalciuria is one of the most frequent metabolic disorders associated with nephrolithiasis and/or nephrocalcinosis leading to Chronic Kidney Disease (CKD) and bone complications in adults.

Hypercalciuria can be secondary to increased intestinal absorption and/or increased renal distal tubular reabsorption of calcium due to increased active vitamin D, i.e. 1,25(OH)2D, levels. The management of hypercalciuria is challenging. Classic management based on hyperhydration and dietary advice has low impact on calciuria and therefore on CKD progression. Other strategies such as hydrochlorothiazide can be proposed, however with an uncertain medical benefit in view of side effects (hypokalemia, asthenia, potential cutaneous long-term side effects).

Azoles are known to inhibit the 1α-hydroxylase and therefore decrease 1,25(OH)2D levels. These antifungal drugs are commonly used in neonates, infants and adults; pharmacokinetic data are well described. Recently, to improve azoles tolerance, fluconazole has been successfully reported to reduce calciuria in patients with CYP24A1 mutation (1 adult) or NPTIIc mutations (1 child), while maintaining a stable renal function. Based on these observations, the investigators hypothesize that fluconazole is effective to decrease and normalize calciuria in patients with hypercalciuria and increased 1,25(OH)2D levels.

The primary objective is to demonstrate that fluconazole normalizes or decreases calciuria after 18 weeks of treatment in patients with hypercalciuria and increased 1,25(OH)2D levels.

The secondary objectives aim to describe:

* the effects of fluconazole on the evolution over time of the calcium/phosphate metabolism,
* the evolution of renal function,
* the cohort at Baseline and after 4 months of treatment period,
* the safety of fluconazole,
* the onset of potential mycological resistances,
* and the treatment compliance. This is a prospective, interventional, national, randomized in 2 parallel groups (1:1), controlled versus placebo, double blind trial.

This study will involve patients between 10 and 60 years of age suffering from nephrolithiasis and/or nephrocalcinosis with hypercalciuria (> 0.1 mmol/kg/d) and increased 1,25 (OH)2D levels (≥ 150 pmol/l) and 25-OH-D levels (≥50 nmol/L).

FLUCOLITH study is a unique opportunity to develop a new indication of a well-known and not expensive drug (e.g. fluconazole) in rare renal diseases, the ultimate objective being the secondary prevention of CKD worsening in these patients.

If the results of this proof-of-concept randomized controlled trial are positive, the investigators will propose an extension phase to evaluate the long term efficacy and safety of fluconazole on renal and bone parameters.

ELIGIBILITY:
Inclusion Criteria:

* Patients who presented in their medical history nephrolithiasis and/or nephrocalcinosis
* Patients who have at inclusion (V1), a local biological evaluation with:

  * 24-hour urine calcium > 0.1 mmol/kg/day,
  * and 1,25(OH)2D levels ≥ 150 pmol/L,
  * and 25-OH-D levels ≥ 20 nmol/L,
  * and calcemia levels ≤ 2.65 mmol/L.
* Children from 10 years
* Adults until 60 years
* Women of child-bearing potential (including sexually active adolescent females) must use highly effective methods of contraception (Annex 7 CTFG recommendations) during the study period. Likewise, partners of male patients of child-bearing potential must use highly effective methods of contraception. Male patients must use condoms.
* Patients insured or beneficiary of a health insurance plan
* Evidence of signed and dated informed consent document(s) indicating that the subject and/or his parents/legal guardian has/have been informed of all pertinent aspects of the trial.

Exclusion Criteria:

* Patient who already received fluconazole or ketoconazole during the last 6 months before inclusion
* Patient weight below than 28 kg
* Patient with BMI >35
* Women menopaused
* Patients who cannot stop hydrochlorothiazide or other diuretics during the screening and study period
* Patients who cannot stop vitamin D supplementation and/or calcium supplementation (drugs, enriched waters, etc.) during the study period
* Hypersensibility to fluconazole and/or other derivative azoles and/or excipients
* Due to the presence of lactose excipient, patients presenting rare hereditary abnormalities of galactose intolerance, of Lapp lactase deficit or of glucose-galactose malabsorption
* Patients who need co-administration with other drugs known to prolong the QT interval and metabolized by cytochrome P450 (CYP) 3A4 (pimozide, quinidine and erythromycin; the exhaustive list of drugs known to prolong the QTc is available on: https://crediblemeds.org).
* Patients with iatrogenic hypercalciuria (vitamin D intoxication, immobilization)
* Relating to the risk of QT interval prolongation:

  1. congenital Long QT syndrome;
  2. familial history of sudden cardiac death before 50 years of age;
  3. cardiopathy: ischemia or myocardial infarction, congestive cardiac insufficiency, left ventricle hypertrophy, cardiomyopathy, conduction trouble within 6 months preceding the inclusion;
  4. arrhythmia history (in particular ventricular arrhythmia, auricular fibrillation or recent rhythm recovery after an auricular fibrillation);
  5. electrolytic instabilities: hypokalemia, hypomagnesemia, hypocalcemia ;
  6. bradycardia (< 50 beats per minute) ;
  7. acute neurological events (i.e. intracranial hemorrhage or sub-arachnoid, cerebrovascular accident, intracranial trauma) within 6 months preceding the inclusion;
  8. adult patients with a QT interval/corrected QT interval > 470ms for women and > 450ms for men at the ECG performed at the inclusion visit (V1). For children from 10 years, the QT interval/corrected QT interval should be > 460ms for girls and > 450ms for boys.
* Children with a history of cardiac pathology
* Patients with an estimated glomerular filtration rate < 60 mL/min/1.73m²
* Patients with a liver disease or an abnormality in the initial liver lab test
* Patients with enuresis
* Patients with another cause of identified lithiasis
* Patients suffering from granulomatosis pathology such as sarcoidosis
* Patient with hyperparathyroidism
* Women who are pregnant or breast feeding, or who have a project of pregnancy before the end of the study
* Patients with a project of travelling in a sunny area during the study period
* Immunodeficient patients
* Patients with other diseases or disorders that could preclude assessment
* Patient who is participating in another research study that may interfere with the results or conclusions of this study
* Patients under judicial protection.

Ages: 10 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-13 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Proportion of patients with normalization of calciuria | Baseline (V1) and 18 weeks of treatment (V7)
  Proportion of patients with normalization of 24-hour calciuria (≤ 0.1 mmol/kg/d) between Baseline (V1) and W18 (V7), or with a relative change of 30% of 24-hour calciuria between Baseline (V1) and W18 (V7) for patients who still have at W18 a 24-hour calciuria> 0.1mmol/kg/d.

SECONDARY OUTCOMES:
Evolution over time of the calcium/phosphate metabolism (serum and urines dosages) | Baseline (V1), 18 weeks of treatment (V7)
  Serum: calcium, ionized calcium, phosphate, magnesium, PTH, 25-OH-D, 1,25(OH)2D, 24-25 (OH)2 D, 25-OH-D:24-25(OH)2D ratio, total alkaline phosphatase.
Serum creatinine | Baseline (V1), 18 weeks of treatment (V7)
  Evolution of renal function
number of lithiasis, nephrocalcinosis | Baseline (V1), 18 weeks of treatment (V7)
  Evolution of renal function
size of lithiasis, nephrocalcinosis | Baseline (V1), 18 weeks of treatment (V7)
  Evolution of renal function
Quantity of calcium intakes | 18 weeks
  Anthropometry
Quantity of sodium intakes | 18 weeks
  Anthropometry
Quantity of protein intakes | 18 weeks
  Anthropometry
bone alkaline phosphatases | 16 weeks
  Bone evaluation with biomarkers
FGF23 | 16 weeks
  Bone evaluation with biomarkers
Klotho | 18 weeks
  Bone evaluation with biomarkers
femoral neck (FN) assessed with Dual energy x-ray absorptiometry (DXA): | at randomization (day 0)
  Bone evaluation with biomarkers
lumbar spine vertebra 2 to 4 (LS2-4) areal bone mineral density assessed with Dual energy x-ray absorptiometry (DXA): | at randomization (day 0)
  Bone evaluation with biomarkers
total body (TB) areal bone mineral density assessed with Dual energy x-ray absorptiometry (DXA): | at randomization (day 0)
  Bone evaluation with biomarkers
Safety evaluation through the study : cardiac evaluation | Baseline (V1)
  Cardiac evaluation : electrocardiogram, corrected QT interval
Safety evaluation through the study : cardiac evaluation | 4 weeks
  Cardiac evaluation : electrocardiogram, corrected QT interval
Safety evaluation through the study : cardiac evaluation | 10 weeks
  Cardiac evaluation : electrocardiogram, corrected QT interval
Safety evaluation through the study : blood analysis | 20 weeks
  Hepatic functions : aspartate transaminase
Safety evaluation through the study : blood analysis | 20 weeks
  Hepatic functions : bilirubin
Safety evaluation through the study : blood analysis | 20 weeks
  Hepatic functions : gamma-glutamyl-transpeptidase
Safety evaluation through the study : blood analysis | 20 weeks
  Lactate dehydrogenase
Safety evaluation through the study : blood analysis | 20 weeks
  phosphoremia
Safety evaluation through the study : blood analysis | 20 weeks
  Calcemia
Safety evaluation through the study : blood analysis | 20 weeks
  Serum creatinine
Safety evaluation through the study : blood analysis | 20 weeks
  Albumin
Safety evaluation through the study : blood analysis | 18 weeks
  Hepatic functions : alanine aminotransferase
Safety evaluation through the study : blood analysis | 20 weeks
  Complete blood cell counts
Proportion of patients that developed mycological resistance | 18 weeks
  Mycological urine samples will be collected to evaluate the onset of potential mycological resistances to Candida. A description of the proportion of patients that developed at least one mycological resistance into the study will be performed by treatment arm, with a listing of the given resistances.
Proportion of patients that developed mycological resistance | 18 weeks
  Mycological buccal samples will be collected to evaluate the onset of potential mycological resistances to Candida. A description of the proportion of patients that developed at least one mycological resistance into the study will be performed by treatment arm, with a listing of the given resistances.
Compliance assessment | every month from Randomization (V2) to 18 weeks of treatment (V7)
  Compliance under treatment (fluconazole or placebo) will be measured by accountability of returned study treatment and information recorded on patients' diary. Level of compliance will be described separately at several follow-up times
Quality of life and treatment satisfaction assessments : adults | The endpoint will be the variation of total score between Randomization (V2) and 18 weeks of treatment (V7)
  Quality of life will be assessed with SF-36 auto-questionnaire (for adult patients)
Quality of life and treatment satisfaction assessments : children and adolescents | The endpoint will be the variation of total score between Randomization (V2) and 18 weeks of treatment (V7)
  PedsQL auto-questionnaire (PedsQL 8-12 years for children, and PedsQL 13-18 years for adolescents).

CONTACTS AND LOCATIONS:
Overall Officials: Aurélia BERTHOLET-THOMAS, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (11):
- France (11):
  - Service de Néphrologie Rhumatologie Dermatologie Pédiatrique, Bron
  - CHU de Dijon, Dijon
  - Hôpital Edouard Herriot, Lyon
  - APHM - CHU Conception, Marseille
  - CHR Metz-Thionville, Metz
  - CHU de Nantes, Nantes
  - Hôpital Universitaire Necker, Paris
  - APHP - Hôpital Européen Georges Pompidou HEGP, Paris
  - Hôpital Universitaire Necker-Enfants Malades, Paris
  - CHU Rennes Pontchaillou, Rennes
  - CHU de Strasbourg, hôpital de Hautepierre, Strasbourg

REFERENCES:
- [Derived] Bertholet-Thomas A, Portefaix A, Flammier S, Dhelens C, Subtil F, Dubourg L, Laudy V, Le Bouar M, Boussaha I, Ndiaye M, Molin A, Lemoine S, Bacchetta J. Fluconazole in hypercalciuric patients with increased 1,25(OH)2D levels: the prospective, randomized, placebo-controlled, double-blind FLUCOLITH trial. Trials. 2022 Jun 16;23(1):499. doi: 10.1186/s13063-022-06302-z. PMID 35710560